CLINICAL TRIAL: NCT02549885
Title: Efficacy of Proprioceptive Neuromuscular Facilitation in Pain Relief in Women With Migraine
Brief Title: Efficacy of Proprioceptive Neuromuscular Facilitation in Pain Relief
Acronym: PNF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, DÉBORA WANDERLEY VILLELA, Master, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ECCR2015
Record Dates: First submitted 2015-09-10; First posted 2015-09-15 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Migraine Disorders
Keywords: Migraine disorders; Muscle stretching exercises
MeSH Terms: conditions — Migraine Disorders | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PNF contract-relax (Experimental): Proprioceptive neuromuscular facilitation, using the technique of contract-relax on neck diagonal.
  Interventions: Other: PNF contract-relax
- Static stretching (Experimental): Static stretching of neck muscles.
  Interventions: Other: Static stretching

INTERVENTIONS:
Other: PNF contract-relax — Proprioceptive neuromuscular facilitation, using the technique of contract-relax on neck diagonal.
  Arms: PNF contract-relax
Other: Static stretching — Static stretching of neck muscles.
  Arms: Static stretching

SUMMARY:
The purpose of this study is to determine whether the contract-relax technique of proprioceptive neuromuscular facilitation, and the static stretching exercise are effective in reducing the frequency, intensity and duration of headache and in improving the perception of quality of life in women with migraine.

DETAILED DESCRIPTION:
This is an randomized clinical trial, double blind, comparing two interventions in women with migraine, whose diagnosis was confirmed by a neurologist.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18and 40 years
* Clinical diagnosis of migraine
* Participants with at least one day with acute migraine per month, with attacks lasting 4-72 hours.

Exclusion Criteria:

* Obesity type I, II or III, according to the classification of Body Mass Index.
* Pregnancy, lactation or both.
* Presence of meningitis, demyelinating diseases, cerebral aneurysm, intracranial hypertension, myopathies, myelopathy, fibromyalgia, symptomatic neck disc herniation, rheumatoid arthritis and history of tumors in the brain or spine.
* Participants who performed other manual therapeutic interventions or other physical therapy modalities in the head or neck during the survey period.
* Participants who have daily prophylactic medication for migraine.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Pain change | "Change from Baseline Pain at 8th - 10th week"; "Change from Baseline Pain at 12th - 14th week"
  "Daily headache"
The global perception of change | "global perception of change at 12th - 14th week"
  "Patient Global Impression of Change Scale"
Feasibility for successful random allocation | "12 months"
  "successful random allocation of 30 patients during a 12-months period"
Proportion of eligible patients randomly assigned for each group (target ≥70%) | "12 months"
  "the proportion of eligible patients randomly assigned for each group (target ≥70%)"
Proportion of eligible patients who completed 30-day follow-up (target ≥95%) | "12 months"
  "the proportion of randomly assigned patients who completed 30-day follow-up after the end of the treatment (target ≥95%)"

SECONDARY OUTCOMES:
Change in Medicine intake in migraine attacks | "Change from Baseline Medicine intake at 8th - 10th week"; "Change from Baseline Medicine intake at 12th - 14th week"
  "Daily headache"
Change in Adverse effects of the intervention | "Change from Baseline adverse effects at 8th - 10th week"; "Change from Baseline adverse effects at 12th - 14th week"
  Daily headache
Change in Neck mobility | "Change from Baseline neck mobility at 8th - 10th week"; "Change from Baseline neck mobility at 12th - 14th week"
  Goniometer "Cervical Range of Motion (CROM)"
Change in pressure pain threshold | "Change from Baseline pressure pain threshold at 8th - 10th week"; "Change from Baseline pressure pain threshold at 12th - 14th week"
  "Computerized Algometer"
Change in neck disability index | "Change from Baseline neck disability index at 8th - 10th week"; "Change from Baseline neck disability index at 12th - 14th week"
  Questionnaire "Neck disability index"
Change in severity of migraine-related disability | "Change from Baseline Migraine disability assessment at 8th - 10th week"; "Change from Baseline Migraine disability assessment at 12th - 14th week"
  Questionnaire "Migraine disability assessment"

CONTACTS AND LOCATIONS:
Overall Officials: DÉBORA W VILLELA, MASTER, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Departamento de Fisioterapia da Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No